CLINICAL TRIAL: NCT03215836
Title: Obesity, Metabolic Dysregulation and the Airway Epithelium in Asthmatics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Jewish Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-2522
Record Dates: First submitted 2017-06-12; First posted 2017-07-12 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Asthma; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Asthma; Obesity; Metabolic Syndrome | interventions — Bronchoscopy

STUDY DESIGN:
Intervention Model Description: This is a cross sectional pilot study comparing specific metabolic pathways in bronchial airway epithelial cells and the nasal epithelium across the following patient groups:
  1. Obese (BMI ≥ 30) asthmatics without metabolic syndrome,
  2. Obese asthmatics with metabolic syndrome,
  3. Obese non-asthmatics, and
  4. Non - obese (lean > 18 <= 25, OW > 25 - <30) asthmatics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Obese Asthmatics (Other): BMI >/= 30 and without metabolic syndrome
  Interventions: Procedure: Bronchoscopy and Nasal Epithelium Brush Sampling
- Obese Astmatics (Other): BMI >/= 30 and with metabolic syndrome
  Interventions: Procedure: Bronchoscopy and Nasal Epithelium Brush Sampling
- Obese non-asthmatics (Other): BMI >/= 30
  Interventions: Procedure: Bronchoscopy and Nasal Epithelium Brush Sampling
- Non - obese asthmatics (Other): BMI: lean > 20; Normal >/= 20 to <25; overweight </= 25 to < 30;
  Interventions: Procedure: Bronchoscopy and Nasal Epithelium Brush Sampling

INTERVENTIONS:
Procedure: Bronchoscopy and Nasal Epithelium Brush Sampling — After meeting screening criteria, participants will undergo further evaluation to determine whether or not inclusion and exclusion criteria are met. Participants will undergo a baseline evaluation, lung function testing and a subsequent bronchoscopy and nasal epithelial brush sampling in those that meet study enrollment.

SUMMARY:
The objective of this pilot study is to determine whether obesity and metabolic syndrome are in fact synergistic in relation to airway nitric oxide (NO) biology. To do so, the investigators want to determine how obesity and the metabolic syndrome relate to metabolism in bronchial airway epithelial cells and the nasal epithelium.

DETAILED DESCRIPTION:
This is a cross sectional pilot study comparing specific metabolic pathways in bronchial airway epithelial cells and the nasal epithelium across the following patient groups:

1. Obese (Body Mass Index (BMI) ≥ 30) asthmatics without metabolic syndrome,
2. Obese asthmatics with metabolic syndrome,
3. Obese non-asthmatics, and
4. Non - obese (lean > 18 <= 25, Overweight (OW) > 25 - <30) asthmatics.

Participants in these groups will be matched by gender, age and asthma severity. To be enrolled, participants must be non-current smokers and be controlled. After meeting screening criteria, participants will undergo further evaluation to determine whether or not inclusion and exclusion criteria are met. Participants will undergo a baseline evaluation, lung function testing and a subsequent bronchoscopy and nasal epithelial brush sampling in those that meet study enrollment.

Participants without a bronchodilator withhold will be scheduled to undergo a methacholine test. Those that qualify will undergo a bronchoscopy to obtain bronchoalveolar lavage and airway epithelial cells and nasal epithelial brush sampling for gene expression studies. After the procedure is done and post bronchoscopy safety standards are met, participants will be discharged from the inpatient Clinical Translational Research Center (CTRC) recovery area. The research coordinator will call the participant on the night of the procedure and on the next day to document post-procedure clinical stability.

ELIGIBILITY:
Inclusion Criteria:

For ALL Groups

1. Adequate completion of informed consent process with written documentation
2. Male and female patients, ≥ 18 - 65 years old
3. Smoking history <10 pack years and no smoking in the last year

   **Subjects can be included in the study if they are on blood pressure treatment and are on a diet control/exercise only treatment of diabetes.
4. Specific to Asthma Groups

i. From all racial/ethnic backgrounds with a diagnosis of asthma based on physician diagnosis for >6 months

1. Specific to Metabolic Syndrome Group. Metabolic syndrome diagnosis based on having at least any three of: a. Triglycerides ≥ 150 mg/dl; b. High-density lipoproteins (HDL) cholesterol ≤ 50 mg/dl for women and ≤ 40 mg/dl for men; c Fasting blood glucose ≥ 100 mg/dl; d. Waist circumference > 40 inches males and > 35 inches females); e. Previously diagnosed hypertension or on antihypertensive medication; f. Blood pressure greater than 130/85 on two consecutive measurements.
2. Specific to Non-Metabolic Syndrome Group a. Baseline pre-bronchodilator forced expiratory volume (FEV1) of 50% or greater of predicted with a 12% or greater bronchodilator (BD) response to 4 puffs of albuterol or PC20 methacholine (16 mg) if no BD response; b. BMI ≥ 30

   Metabolic syndrome diagnosis based on having at least any three of:

   i. Triglycerides ≥ 150 mg/dl; ii. HDL cholesterol ≤ 50 mg/dl for women and ≤ 40 mg/dl for men; iii. Fasting blood glucose ≥ 100 mg/dl; iv. Waist circumference > 40 inches males and > 35 inches females); v. Previously diagnosed hypertension or on antihypertensive medication; vi. Blood pressure greater than 130/85 on two consecutive measurements.
3. Specific to Non-Obese Group a. Body Mass Index (BMI) < 30

   b. Specific to Non-Asthma Group i. No history of asthma or any other airway diseases; ii. Pulmonary function test within normal limits; iii. BMI ≥ 30.

Exclusion Criteria (all groups):

1. Significant or uncontrolled concomitant medical illness (PI discretion) including, but not limited to heart disease, cancer, diabetes (HbAc1 > 6.5), renal disease (creatinine > 2.0) at Visit 0, neurological (brain damage) or psychiatric disorder (diagnosed by a mental health professional of behavioral or mental pattern that may cause suffering or a poor ability to function in life);
2. Chronic renal failure (creatinine > 2.0) at screening (associated with higher asymmetric dimethylarginine (ADMA) levels);
3. Current statins use (statins lower ADMA levels);
4. On diabetic medications;
5. Positive pregnancy test;
6. Positive urine cotinine and/or urine tetrahydrocannabinol (THC) test;
7. Current or recent (within 30 days) investigational treatment or participation in another interventional research study (including non-pharmacologic interventions);
8. Unable or unlikely to complete study assessments or the study intervention (i.e. bronchoscopy) poses undue risk to patient in the opinion of the investigator.

   a. Specific to Asthma Groups i. Respiratory tract infection within the last 4 weeks; ii. Oral or systemic corticosteroids (CS) burst within the last 4 weeks; iii. Asthma-related hospitalization within the last 2 months; iv. Asthma-related ER visit within the previous 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08-10 (Actual); Primary Completion 2027-03-10 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of L-arginine-NO biosynthesis pathways in the airway epithelium in obese and non-asthmatics. | Within 6 months of collection
  L-arginine-NO biosynthesis pathways will be measured in the airway epithelium of mild to moderate controlled obese and non-obese asthmatics with metabolic syndrome by ELISA and western blot analysis.
Measurement of oxidative stress in the airway epithelium in obese and non-asthmatics. | Within 6 months of collection
  Oxidative stress will be measured in the airway epithelium of mild to moderate controlled obese and non-obese asthmatics without metabolic syndrome by Griess Reaction and western blot analysis.

SECONDARY OUTCOMES:
Measurement of mitochondrial density | Within 6 months of collection
  Mitochondrial density will be measured from cells obtained by one time pulmonary lavage during bronchoscopy.
Measurement of mitochondrial structural differences. | Within 6 months of collection
  Mitochondrial structural differences will be measured from cells obtained by one time pulmonary lavage during bronchoscopy.
Patterns of Gene expression found in the nasal epithelium. | Within 6 months of collection
  Nasal epithelial cells will be obtained by one time nasal brushings and gene expression patterns will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Holguin, MD, MPH, Principal Investigator — University of Colorado Denver, Anschutz Medical Campus
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
Airway epithelial cells, serum samples and bronchoalveolar lavage (BAL) fluid and BAL cells being collected under this protocol will be collected in UC Denver and sent to National Jewish Hospital (NJH) as per agreed protocols. Specimens/instruments will be completely de-identified and the only data that will be sent to Hong Wei Chu's lab at National Jewish Hospital (NJH) will be specimens labeled with a code.